CLINICAL TRIAL: NCT04440605
Title: A Study to Confirm the Accuracy of Locally Advanced Gastric Cancer Diagnosis: A Prospective, Multicenter, Cohort Study
Brief Title: A Study to Confirm the Accuracy of Locally Advanced Gastric Cancer Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: RenJi Hospital (Other); Ruijin Hospital (Other); West China Hospital (Other); Beijing 302 Hospital (Other); Fudan University (Other); Peking University International Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Fujian Medical University Union Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Chinese PLA General Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Tianjin Medical University General Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Peking University People's Hospital (Other); Weifang People's Hospital (Other); Second Hospital of Jilin University (Other); Fujian Province Tumor Hospital (Other); Shanxi Province Cancer Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Shanghai Zhongshan Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital of Xiamen University (Other); Beijing Hospital (Other Government); Beijing Friendship Hospital (Other); Qingdao Municipal Hospital (Other); Guangdong Provincial People's Hospital (Other); Affiliated Hospital of Qinghai University (Other); Shandong Provincial Hospital (Other Government); The First Hospital of Jilin University (Other); Nanfang Hospital, Southern Medical University (Other); Zhongshan Hospital Xiamen University (Other); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Ziyu Li, MD, M.D., Ph.D., Peking University
Other Study IDs: 2019YJZ55
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Gastric Cancer; Gastric Cancer Stage; CT; Neoadjuvant Therapy
Keywords: Gastric cancer; Clinical TNM staging; Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adenocarcinoma tissue sample retrieved by endoscopic and sugical methods
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cI: clincal TNM stage I
  Interventions: Procedure: Preoperative staging--D2 gastrectomy--Postoperative staging
- cII: clinical TNM stage II
  Interventions: Procedure: Preoperative staging--D2 gastrectomy--Postoperative staging
- cIII: clinical TNM stage III
  Interventions: Procedure: Preoperative staging--D2 gastrectomy--Postoperative staging

INTERVENTIONS:
Procedure: Preoperative staging--D2 gastrectomy--Postoperative staging — Preoperative TNM staging under CT scan plus endoscopy endoscopic biopsy, and postoperative staging after D2 gastrectomy

SUMMARY:
With the introducing of neoadjuvant therapy, it becomes ever more important to evaluate the preoperative TNM (cTNM) stage accurately facilitating preoperative treatment as well as the adjuvant therapy.

At present, the recommendation of neoadjuvant chemotherapy varies among guidelines especially between eastern and western countries. According to the updated Japanese gastric cancer treatment guidelines (ver.5), neoadjuvant chemotherapy is the recommended standard procedure for patients with cT2-4 stages. However, the acknowledgement of preoperative therapy accompanied by the higher risk of overtreatment. As mentioned in JCOG1302-A, the overall precision rate in cT staging is 38.8%. Patients diagnosed with pI stages postoperatively account for 6.5% in cT3-4N+ treatment indicating more likely to avoiding the overtreatment comparing to patients with other cT stages.

Inspired by JCOG1302-A, this multicentre study prospectively collect data in preoperative TNM staging assessment using CT(computed tomography, CT) scan and the postoperative TNM (pTNM) staging according to histopathologically examination. By analyzing the accordance between the cTNM and pTNM, this study aims to evaluate the current accuracy of the cTNM staging in china, verifying the proportion of pI stages less than 5% in cIII stage diagnosis patients, learning the overtreating rate in neoadjuvant chemotherapy in China and furthermore, to discover the scope of beneficiaries for neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Confirm the inclusion of pathological stage I (pI) among clinical stage III(T3-4aNx) (cIII) diagnosis patients less than 5% II. Figure out the suitable criterion of NAC and avoid overtreatment, by examining the rate of pI rate in different diagnostic criterion groups, including cIII, TxNy(x+y>4), cN1-3, cT3-4.

III. Evaluate the current state of diagnostic accuracy of preoperative CT staging in china.

OUTLINE:

This is a prospective, multi-centers, cohort study of clinical TNM staging diagnostic accuracy.

Patients are divided into 3 preoperative stage groups according to AJCC 8th edition (cI, cII, cIII) preoperatively. All patients receive the D2 gastrectomy after cTNM diagnosis and the pathological stages is given following surgery.

The concordance of preoperative staging is evaluated in each cohorts as well as the subgroups to obtain the accuracy rate. The pI proportion will calculate in each latent criterion groups to assess the suitable NAC criteria.

PROJECTED ACCRUAL: A total of 968 patients will be accrued for this study within two years.

ELIGIBILITY:
Inclusion Criteria:

* Histological prove of adenocarcinoma of the stomach by endoscopy
* Preoperative imaging data by contrast-enhanced CT and clinical TNM stages were given
* No evidence of stage IV disease
* No previous gastrectomy or preoperative treatment.

Exclusion Criteria:

* Discovery of distant metastasis (stage IV) during surgery
* Number of retrieved lymph node less than 15

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with endoscopically biopsy-proven adenocarcinoma of the stomach and with contrast-enhanced CT cI-III diagnosis prior to surgery will receive treatment.
Sampling Method: Probability Sample
Enrollment: 968 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of cIII | 1.5 years
  Proportion of pathological stage I among clinical stage III(T3-4aNx) diagnosis patients

SECONDARY OUTCOMES:
Diagnostic Accuracy of cTxNy | 1.5 years
  Proportion of pathological stage I among clinical TxNy(x+y>4) stage diagnosis patients
Diagnostic Accuracy of cN+ | 1.5 years
  Proportion of pathological stage I among clinical N1-3 stage diagnosis patients
Diagnostic Accuracy of cT3/4 | 1.5 years
  Proportion of pathological stage I among clinical T3-4 stage diagnosis patients
Diagnostic Accuracy of cTN | 1.5 years
  The concordance rate for clinical staging

CONTACTS AND LOCATIONS:
Locations (38):
- China (38):
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - 301 Hospital, Beijing, Beijing Municipality
  - 302 Military Hospital of China, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Tumor Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital of Xiamen University, Xiamen, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangdong Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Heilongjiang Cancer Hospital, Harbin, Heilongjiang
  - Wuhan Union Hospital, Wuhan, Hubei
  - Jiangsu People's Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital-Dalian Medical University, Dalian, Liaoning
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Fudan University Cancer center, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Renji Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanxi Tumour Hospital, Taiyuan, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

REFERENCES:
- [Background] Fukagawa T, Katai H, Mizusawa J, Nakamura K, Sano T, Terashima M, Ito S, Yoshikawa T, Fukushima N, Kawachi Y, Kinoshita T, Kimura Y, Yabusaki H, Nishida Y, Iwasaki Y, Lee SW, Yasuda T, Sasako M; Stomach Cancer Study Group of the Japan Clinical Oncology Group. A prospective multi-institutional validity study to evaluate the accuracy of clinical diagnosis of pathological stage III gastric cancer (JCOG1302A). Gastric Cancer. 2018 Jan;21(1):68-73. doi: 10.1007/s10120-017-0701-1. Epub 2017 Feb 13. PMID 28194522